CLINICAL TRIAL: NCT01266824
Title: Randomized Control Trial of the Effects of Proparacaine on the Pain Response to Mydriatic Eye Drops
Brief Title: Proparacaine and Mydriatic Eye Drops
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment for the study has been terminated due to poor enrollment
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Amy M Cohen, MD, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 812311
Record Dates: First submitted 2010-12-21; First posted 2010-12-24 (Estimated); Results first posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-02

CONDITIONS: Pain; Retinopathy of Prematurity
Keywords: Pain; Retinopathy of Prematurity; Neonates
MeSH Terms: conditions — Pain; Retinopathy of Prematurity

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Proparacaine (Experimental): Infants in this group will receive 1 drop of Proparacaine Hydrochloride Ophthalmic Solution (anesthetic eye drop) into each eye prior to receiving mydriatic eye drops
  Interventions: Drug: Proparacaine Hydrochloride Ophthalmic Solution
- Standard of Care (No Intervention): Infants in this arm will not receive Proparacaine Hydrochloride Ophthalmic Solution (anesthetic eye drop) prior to mydriatic eye drops.

INTERVENTIONS:
Drug: Proparacaine Hydrochloride Ophthalmic Solution — 1 drop into each eye once prior to the first set of mydriatic (dilating) eye drops
  Arms: Proparacaine

SUMMARY:
In this study, we will be evaluating whether premedication with an anesthetic eye drops leads to a decreased sensation of pain when given dilating eye drops prior to eye examinations to evaluate for retinopathy of prematurity in neonatal intensive care unit (NICU) infants.

DETAILED DESCRIPTION:
A. Randomization of subjects: Infants will be randomized to receive Proparacaine versus no intervention based on computerized randomization performed by our statistician. Due to the lack of a placebo group, practitioners present at the time of examination will not able to be blinded to group assignment. Each infant will only be enrolled for one examination.

B. Monitor setup/application: The Central Nervous System (CNS) Neonatal Neurological Monitor (Moberg Research) will be used to videotape each patient encounter and record vital sign information during the study period. The CNS monitor will record physiologic variables indirectly via cables attached to the bedside monitor. Before scheduled eye drop administration takes place, the appropriate connections between the bedside monitor and CNS monitor will be made in order to continuously record heart rate, respiratory rate, pulse oximetry, and blood pressure. A video camera attached to the CNS monitor will also be positioned to capture the subjects' facial activity and gross body movements. The monitor will be set up with enough time prior to eye drop administration such that baseline data can be collected before any intervention is performed. In addition, a video recording of the method of eyedrop administration will be assessed. The monitor will remain in place up to 5 minutes after completion of eye drop administration.

C. Eye drop administration: The CNS Monitor will be in place at least 3 minutes prior to administration of any eye drops to record baseline data on the infant. One drop of Proparacaine anesthetic ophthalmic solution will be applied to each eye of infants randomized to receive Proparacaine prior to the mydriatic eye drops. At least 30 seconds and no longer than 5 minutes after administration of Proparacaine, the mydriatic eye drops will be given as per routine standard practice for ophthalmologic examinations in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Infants admitted to the Pennsylvania Hospital NICU who require an ophthalmologic examination.

Exclusion Criteria:

* Infants with congenital anomalies, seizures, or other neurologic conditions or malformations that may alter the pain response
* Infants with corneal abrasions, corneal ulcers or other relative or absolute contraindications to proparacaine administration

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy MP Cohen, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Pennsylvania Hospital NICU, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study was terminated due to poor enrollment.
Groups:
- Proparacaine: Infants in this group will receive 1 drop of Proparacaine (anesthetic eye drop) into each eye prior to receiving mydriatic eye drops
  Proparacaine Hydrochloride Ophthalmic Solution : 1 drop into each eye once prior to the first set of mydriatic (dilating) eye drops
- Standard of Care: Infants in this arm will not receive Proparacaine (anesthetic eye drop) prior to mydriatic eye drops.
Period: Overall Study
Arm/Group | Proparacaine | Standard of Care
Started | 2 | 3
Completed | 0 | 0
Not Completed | 2 | 3
Not completed — Study terminated prior to completion | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proparacaine | Standard of Care | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.14 (0.028) | 0.12 (0.006) | 0.13 (0.016)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in PIPP Score
Description: Comparison of the change in Premature Infant Pain Profile (PIPP) scores from baseline to the time immediately following mydriatic drop administration between the groups of infants who do and do not receive Proparacaine eye drops prior to mydriatic drops. The PIPP score is a scale to determined pain response that was designed for use in preterm and term infants. It is based on both physiologic and behavioral changes exhibited by infants during the study period of 30s (facial changes, HR, O2 saturation). There are correction factors for gestational age and baseline state at time of scoring. Scores can range from 0-21 with the maximum score dependent on the infant's gestational age. A score >7 typically indicates a pain response while a score >12 indicates more severe pain.
Time Frame: Change from baseline to time immediately following mydriatic drop administration
Population: Due to poor enrollment, this study was not completed and no patients were analyzed as a part of the randomized controlled trial.
Arm/Group | Proparacaine | Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: PIPP Score
Description: PIPP scores measure immediately after Proparacaine administration
Time Frame: within 5 minutes after Proparacaine administration
Population: as for outcome 1
Arm/Group | Proparacaine | Standard of Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Bradycardia/Desaturation
Description: Number of episodes of bradycardia (HR 90) and significant desaturation (event requiring stimulation, per Neonatal Intensive Care Unit (NICU) protocol, to resolve) occurring after the administration of mydriatic and proparacaine eye drops
Time Frame: Within 5 minutes after Proparacaine/mydriatic drop administration until study monitor disconnected
Population: as for outcome 1
Arm/Group | Proparacaine | Standard of Care
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: PIPP Score
Description: PIPP score measure immediately following mydriatic drop administration
Time Frame: within 5 minutes after Mydriatic drop administration
Population: as for outcome 1
Arm/Group | Proparacaine | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Proparacaine | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

LIMITATIONS AND CAVEATS:
Enrollment for the randomized controlled study above was poor and the study was terminated without patient analysis. An observational study of the pain response to mydriatic eye drops without use of Proparacaine was completed in place of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes